CLINICAL TRIAL: NCT03467490
Title: Assessing a Self-care Management Program for Dry Eye Disease Patients Using the Health Educational Intervention Questionnaire
Brief Title: Self-care Management Program for Dry Eye Disease Patients Using the heiQ
Acronym: heiQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 109377
Record Dates: First submitted 2018-02-28; First posted 2018-03-16 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2019-05

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 65 participants will be invited to receive a one-day educational intervention (first study visit) at the Ivey Eye Institute. The educational intervention includes watching a short video series and receiving educational handouts which summarize the content of the videos. Participants will have access to the educational handbook for reference. At two months post-intervention, participants will be invited back to St. Joseph's Hospital to complete the second administration of the heiQ and OSDI. Participants will have an opportunity to ask the ophthalmologist any question during the question and answer period. Participants will then be asked to provide feedback on the video series using a participation satisfaction survey and will be given an educational handbook which may be used to as a reference/guide on how to self-manage
  Interventions: Behavioral: DED self-management
- Control (No Intervention): Patients will continue with treatment as usual without any educational intervention. They will complete the heiQ and OSDI at baseline and 2 months later during a routine office visit. At the 2-month visit, participants will be asked to complete the second administration of the heiQ and OSDI before being offered the opportunity to view the videos series, receive the educational handbook, and provide feedback on the educational material.

INTERVENTIONS:
Behavioral: DED self-management — This an educational intervention. The interventional will include watching a series of short videos and a DED handbook. The short videos will address the following topics: anatomy of the eye, pathophysiology of DED, treatment options for DED, management of DED with allergies/glaucoma/ computer use, and new developments in treatment and research of dry eye disease. The handbook will include tools and resources for self management of DED.
  Arms: Treatment

SUMMARY:
Dry Eye Disease (DED)is a chronic disease without a cure. Empowering patients to engage in better self-care requires knowledge of their disease and skills in self-management, which can lead to improved well-being and quality of life. The Investigation team has developed a DED self-management program (video series and educational booklet) that can be easily implemented into clinical use. The Investigators are going to use the Ocular Surface Disease Index (OSDI) to measure the dry eye in the participants. In addition, the research team plans to use the heiQ (validated questionnaire that assesses self-management and health education programs) to evaluate the DED self-management program by comparing results taken at baseline to 2 months after undergoing the self-management program.

DETAILED DESCRIPTION:
The aim of this study is to assess a self-care management program for dry eye disease (DED) patients using the Health Educational Intervention Questionnaire (heiQ). The heiQ is tool that facilitates a comprehensive evaluation of patient education and self- management interventions for patients with chronic conditions.

Dry Eye Disease is a chronic and may be a progressive condition. Currently, there is no gold standard in the diagnosis or treatment of dry eye disease, but several management options are available. Just like other chronic conditions like diabetes, patients with dry eye must engage in disease modifying behaviours and perform self-care measures, in addition to taking pharmaceutical agents. Patient education is the foundation of an effective management plan.

Various educational programs have been developed in the past for chronic diseases like psoriasis, diabetes, and cardiovascular disease. However, there are limited studies evaluating self-management and educational interventions for patients with ocular diseases or DED. This research team has developed a program to educate patients on self-management of DED. The educational component of the intervention includes a series of short videos and a self-care handbook. Both the video series and handbook include topics ranging from the causes of DED, basic anatomy of the eye, and self-care skills to manage DED symptoms in various environments, such as the work environment and seasonal changes. This intervention aims to deliver useful information about DED, increase patient knowledge and awareness of strategies to reduce and manage symptoms of DED.

The research team will administer two questionnaires at two different time points to all participants-once at baseline and once at two months post-intervention. The first questionnaire is the Ocular Surface Disease Index (OSDI). This questionnaire is used to determine the severity of dry eye symptoms. The second questionnaire is the Health Educational Impact Questionnaire (heiQ). The heiQ is a validated instrument for health education and self-management programs of chronic diseases. It is comprised of 40 questions that represent 8 independent domains. Those domains include: Health-directed activity, Positive and active engagement in life, Self-monitoring and insight, Constructive attitudes and approaches, Skill and technique acquisition, Social integration and support, Health service navigation, and Emotional distress. Results from the heiQ will serve to provide evidence as to whether this educational intervention is effective and should be placed in clinical practice.

Potential participants will be recruited through Dr. Mather's clinical practice at the Ivey Eye Institute at St. Josephs's Hospital London, ON. A Letter of Information (LOI) and an Invitation Poster will be mailed to potential participants. There will be approximately 130 participants recruited from Dr. Mather's Clinic at the Ivey Eye Institute. The participants will be randomly assigned to the treatment arm or the controlled arm. The intervention in total will take up to 4 hours (2 hours in both sessions). In the first session (baseline) following the consent the first heiQ and OSDI will be completed by all the participants. The treatment group (65 participants) will watch a series of educational videos and will leave the baseline session with a DED handbook. The treatment group will agree not to share information from the session and the DED handbook with anyone until after session two. During the second session (2- months post intervention) all the participants will be asked to come back to St. Joseph's hospital to complete the second heiQ and OSDI. At this session all participants will be invited to watch the educational videos. All participants will be provided a DED handbook and all the participants will be asked to complete a feedback survey that will be provided. No data will be collected after the administration of the second set of questionnaires. Participants that have questions if any will have the opportunity to ask the ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

- Participants will be considered eligible for inclusion in the study if they are:

1. moderate to severe dry eye disease patients (have a minimum score of 20 on the Ocular Surface Disease Index and minimum score of 5 on the Canadian Dry Eye Assessment)
2. at least 18 years of age
3. capable of communicating in English 4) willing and able to receive the educational intervention

5) willing and able to conduct DED self-care at home as needed

Exclusion Criteria:

Participants will be considered ineligible for participation in the study if any of the following criteria are met:

1. They are currently participating in other similar studies
2. They are currently undergoing or have undergone any type of self-care management/educational program for dry eye disease
3. unable/unwilling to receive the educational intervention and complete the two administrations of the heiQ 4 ) Unable to communicate fluently in English as the videos and the heiQ survey are both only available in English.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-11-24 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change score in heiQ subscales | 2 months
  Mean change in scores of each of the eight heiQ subscales from baseline to 2-months post-intervention for each arm of the study

SECONDARY OUTCOMES:
Mean Change scores in OSDI scores | 2 Months
  Mean change in scores of OSDI from baseline to 2 month post-intervention for each arm of the study
Mean change score in heiQ subscale 1:Health-directed activity | 2 months
  mean change score in the heiQ subscale 1 (Health-directed activity) from baseline to 2-months post intervention for each arm of the study
Mean change score in heiQ subscale 1: Health-Directed activity | 2 months
  Mean change score in the heiQ subscale 1 (Health-directed activity) from baseline to 2- month post intervention for each individual participant
Mean change score in heiQ subscale 2: Positive and active engagement in life | 2 months
  Mean change score in heiQ subscale 2 (Positive and active engagement in life) from baseline to 2-months post-intervention for each arm of the study
Mean change score in heiQ subscale 2: Positive and active engagement in life | 2 months
  Mean change score in the heiQ subscale 2 (Positive and active engagement in life) from baseline to 2-months post-intervention for each individual participant
Mean change score in heiQ subscale 3: Self-monitoring and insight | 2 months
  Mean change score in the heiQ subscale 3 (Self-monitoring and insight) from baseline to 2-months post-intervention for each arm of the study
Mean change score in heiQ subscale 3: Self-monitoring and insight | 2 months
  Mean change score in the heiQ subscale 3 (Self-monitoring and insight) from baseline to 2-months post-intervention for each individual participants
Mean change score in heiQ subscale 4: Constructive attitudes and approaches | 2 months
  Mean change score in the heiQ subscale 4 (Constructive attitudes and approaches) from baseline to 2-months post-intervention for each arm of the study
Mean change score in heiQ subscale 4: Constructive attitudes and approaches | 2 months
  Mean change score in the heiQ subscale 4 (Constructive attitudes and approaches) from baseline to 2-months post-intervention for each individual participant
Mean change score in heiQ subscale 5: Skill and technique acquisition | 2 months
  Mean change score in the heiQ subscale 5 (Skill and technique acquisition) from baseline to 2-months post-intervention for each arm of the study
Mean change score in heiQ subscale 5: Skill and technique acquisition | 2 months
  Mean change score in the heiQ subscale 5 (Skill and technique acquisition) from baseline to 2-months post-intervention for each individual participant
Mean change score in heiQ subscale 6: Social integration and support | 2 months
  Mean change score in the heiQ subscale 6 (Social integration and support) from baseline to 2 months post intervention for each arm of the study
Mean change score in heiQ subscale 6: Social integration and support | 2 months
  Mean change score in heiQ subscale 6 (Social integration and support) from baseline to 2 months post intervention for each individual participant
Mean change score in the heiQ subscale 7: Health service navigation | 2 months
  Mean change score in heiQ subscale 7 ( Health service navigation) from baseline to 2-months post-intervention for each arm of the study
Mean change score in the heiQ subscale 7: Health service navigation | 2 months
  Mean change score in heiQ subscale 7 ( Health service navigation) from baseline to 2-months post-intervention for each individual participant
Mean change score in heiQ subscale 8: Emotional distress | 2 months
  Mean change score in heiQ subscale 8 (Emotional Distress) from baseline to 2-months post intervention for each arm of the study
Mean change score in heiQ subscale 8: Emotional distress | 2 months
  Mean change score in heiQ subscale 8 (Emotional Distress) from baseline to 2-months post intervention for each individual participant

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided